CLINICAL TRIAL: NCT03426826
Title: Dynamics of Gut Microbiomes in Autism Spectrum Disorder (ASD) Symptoms
Brief Title: The Gut-Brain Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sonia Michail, MD, Physician /Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHLA-18-00065
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder (ASD); Gastro-Intestinal Disorder
Keywords: FMT; Gut Microbiome; Fecal Microbiata Transplantation; Autism Spectrum Disorder; 16s rRNA; Gastro-Intestinal Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Digestive System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Placebo Comparator): Placebo Comparator placebo into the jejunum through upper endoscopy.
  Interventions: Biological: FMT versus placebo
- Arm 2 (Active Comparator): Active Comparator: Donor Stool Transplant Arm 2 will get FMT (Fecal Microbial Transplant) with Healthy Donor Stool into the jejunum through upper endoscopy.
  Interventions: Biological: FMT versus placebo

INTERVENTIONS:
Biological: FMT versus placebo — Biological/Vaccine: Fecal Microbial Transplant versus placebo Fecal Transplant via endoscopy.
  Other Names:
  FMT
  Other Names: fecal microbial transplant vs placebo

SUMMARY:
The purpose of this study is to find out if transplant of fecal matter (stool), also known as fecal microbiota transplantation (FMT), from a healthy person into the intestines of children and young adults with Autism Spectrum Disorder (ASD).

For this study children between the ages of 5-17years will be recruited over 2 years. Children will be recruited who receive an ASD diagnosis using the gold-standard Autism Diagnosis Observation Schedule -2 (ADOS-2) using module 1, 2 or 3 (none, limited or no moderate expressive language). Children diagnosed with these modules of the ADOS-2 may be at greater risk for GI disorders and rigid-compulsive behaviors. Additional assessment of rigid-compulsive behaviors and social communication will be done using the Repetitive Behavioral Scales-Revised (RBS-R) and Social Responsiveness Scale-2 (SRS-2), respectively. KBIT (the Kaufman Brief Intelligence Test) is used at baseline to obtain patient IQ. Total evaluation time is approximately 90 minutes. Following baseline symptom evaluation, a medical exam will be performed to determine whether each child is expressing specific GI symptoms. In addition, parents will fill out the Questionnaire for Pediatric Gastrointestinal Symptoms- Rome III (QPGS-III). Once an ASD diagnosis is confirmed, FMT treatment will be initiated, which typically occurs within 4-6 weeks of the initial diagnosis. Half 50% of the children (n=5) will receive the equivalent of 50 g of stools from a healthy donor into the jejunum through upper endoscopy and the other 50% off children (n=5) will receive Saline solution as Placebo control through upper endoscopy.

Subjects will have a total of 5 visits within 24 weeks including phone call follow up on Day 7 after FMT.

DETAILED DESCRIPTION:
Nearly 1 in 60 children are diagnosed with ASD, a dramatic increase from the start of the 21st century. Although most children with ASD exhibit core social communication deficits, very limited interests, repetitive behaviors and sensory problems, the severity of symptoms and how well each child responds to standard behavioral therapies can vary tremendously from patient to patient. This makes it difficult to enact effective interventions. Other variables also influence the outcomes for ASD patients, including age at first diagnosis, access to care, the quality of treatments and the expertise of interventionists.

Children with ASD also have medical disturbances, which affects their quality of life and compliance in intervention programs. For example, approximately 40 percent of children with ASD have gastrointestinal disturbances (GIDs). Genetics plays a substantial role in risk, but scientists also have determined that non-heritable factors can trigger the expression and severity of ASD symptoms. Clinical research studies from PI laboratories have focused on the gut-brain link that influences ASD symptoms, how a child functions and even responds to interventions .

The investigators hypothesize that children with ASD will tolerate single endoscopic delivery of fecal transplant therapy which will modify their gut microbial profile leading to reduction of repetitive and rigid-compulsive behaviors, based on the Repetitive Behavioral Scales-Revised (RBS-R). Secondary outcomes include improved score in social responsiveness scale and gastrointestinal symptoms . Investigators propose a phase I safety study for the use of FMT in children with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5-17 who have been diagnosed with non-syndromic ASD-s
* Needs upper GI endoscopy
* Clinical Assessment of ASD
* ADOS validated diagnoses of ASD
* Questionnaires: RBS-2 , KBIT, SRS, Rome III Version (QPGS- RIII), Ped QL, SSP

Exclusion Criteria:

* Subjects able to give consent/assent but unwilling to give informed consent/assent
* Prematurity (<36 weeks)
* Pregnancy: testing will be done on FMT day 0 for subjects with childbearing potential
* Subjects with significant renal and liver dysfunction (creatinine > 2 mg/dl and direct bilirubin > 2 mg/dl)
* Subjects with congenital or acquired immunodeficiency, or who are immunosuppressed such as neoplastic disease or organ transplantation), have received or are receiving chemotherapy, or have been diagnosed with HIV.
* Subjects with syndromic disorders of defined genetic cause, and subjects who have severe sensory or motor problems (for example, blindness, deafness, seizures, cerebral palsy)
* Subjects with severe food allergies

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures, safety and tolerability | 24 weeks
  The primary Outcome is safety of FMT and also it is measured by any symptom changes in obsessive/compulsive and repetitive behaviors using the RBS-R questionnaire.

SECONDARY OUTCOMES:
Secondary Outcome Measures, symptom improvement | 24 weeks
  Secondary endpoints will include cognitive improvement using language use in a 10 minute interactive session, Social Responsiveness Scale-2. The SRS-2 is newly available (Western Psychological Services). It is a parent 65-item questionnaire that provides a continuous quantitative measure of three DSM domains, including social behavior, communication, and restricted and repetitive behaviors, normed in typically developing (T-score=50, sd=10) and ASD populations. The SRS-2 offers new DSM-5 subscales. The SRS is used in a variety of clinical and research settings. T-scores of 65 correlate highly with an ASD diagnosis, but do not substitute for the ADOS. Changes in SRS T-scores have been used as a measure of social behavior change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — Children's Hospital Los Angeles; Pat Levitt, Ph.D, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- [Background] Luna RA, Oezguen N, Balderas M, Venkatachalam A, Runge JK, Versalovic J, Veenstra-VanderWeele J, Anderson GM, Savidge T, Williams KC. Distinct Microbiome-Neuroimmune Signatures Correlate With Functional Abdominal Pain in Children With Autism Spectrum Disorder. Cell Mol Gastroenterol Hepatol. 2016 Dec 11;3(2):218-230. doi: 10.1016/j.jcmgh.2016.11.008. eCollection 2017 Mar. PMID 28275689
- [Background] Gorrindo P, Williams KC, Lee EB, Walker LS, McGrew SG, Levitt P. Gastrointestinal dysfunction in autism: parental report, clinical evaluation, and associated factors. Autism Res. 2012 Apr;5(2):101-8. doi: 10.1002/aur.237. PMID 22511450
- [Background] Gorrindo P, Lane CJ, Lee EB, McLaughlin B, Levitt P. Enrichment of elevated plasma F2t-isoprostane levels in individuals with autism who are stratified by presence of gastrointestinal dysfunction. PLoS One. 2013 Jul 3;8(7):e68444. doi: 10.1371/journal.pone.0068444. Print 2013. PMID 23844202
- [Background] Yao MD, von Rosenvinge EC, Groden C, Mannon PJ. Multiple endoscopic biopsies in research subjects: safety results from a National Institutes of Health series. Gastrointest Endosc. 2009 Apr;69(4):906-10. doi: 10.1016/j.gie.2008.05.015. Epub 2009 Jan 10. PMID 19136110
- [Background] Hamilton MJ, Weingarden AR, Sadowsky MJ, Khoruts A. Standardized frozen preparation for transplantation of fecal microbiota for recurrent Clostridium difficile infection. Am J Gastroenterol. 2012 May;107(5):761-7. doi: 10.1038/ajg.2011.482. Epub 2012 Jan 31. PMID 22290405
- [Background] Finegold SM. Therapy and epidemiology of autism--clostridial spores as key elements. Med Hypotheses. 2008;70(3):508-11. doi: 10.1016/j.mehy.2007.07.019. Epub 2007 Sep 29. PMID 17904761
- [Background] Finegold SM. State of the art; microbiology in health and disease. Intestinal bacterial flora in autism. Anaerobe. 2011 Dec;17(6):367-8. doi: 10.1016/j.anaerobe.2011.03.007. Epub 2011 Apr 16. PMID 21524713